CLINICAL TRIAL: NCT01830231
Title: A Randomised Phase II/III Study of Cabazitaxel Versus Vinflunine in Metastatic or Locally Advanced Transitional Cell Carcinoma of the Urothelium
Brief Title: Cabazitaxel vs. Vinflunine in Metastatic or Locally Advanced Transitional Cell Carcinoma of the Urothelium (TCCU)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associació per a la Recerca Oncologica, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Secavin-12
Record Dates: First submitted 2013-04-02; First posted 2013-04-12 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Urothelium Transitional Cell Carcinoma
Keywords: TCCU; Vinflunine; Cabazitaxel; Metastatic; Locally advance
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cabazitaxel; vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabazitaxel (Experimental): Cabazitaxel 25 mg/m2 q3w. Cabazitaxel will be given intravenously once every 21 days, starting at a dose of 25 mg/m2 as a 1-hour intravenous infusion
  Interventions: Drug: Cabazitaxel
- Vinflunine (Active Comparator): • Vinflunine will be given intravenously once every 21 days, starting at a dose of:
  * 320 mg/m2 in patients aged ≤75 years with PS 0 and no prior pelvic radiation
  * 280 mg/m2 in patients aged >75 - ≤80 years, and/or with PS 1 and/or prior pelvic radiation,
  * 250 mg/m2 in patients aged >80 years.
  Interventions: Drug: Vinflunine

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel, to be given intravenously once every 21 days, starting at a dose of 25 mg/m2 as a 1-hour intravenous infusion.
  Other Names: Jevtana
  Arms: Cabazitaxel
Drug: Vinflunine — Vinflunine, to be given intravenously once every 21 days, as a 20 minute intravenous infusion, starting at a dose of:
  * 320 mg/m2 in patients aged ≤75 years with PS 0 and no prior pelvic radiation, and of
  * 280 mg/m2 in patients aged >75 - ≤80 years or with PS 1 or prior pelvic radiation,
  * 250 mg/m2 in patients aged >80 years.
  Other Names: Javlor
  Arms: Vinflunine

SUMMARY:
Due to limited experience with cabazitaxel in TCCU, the study will be started as a randomised phase II study. The aim of the phase II study is to evaluate if the response rates (CR + PR) are sufficiently high to further study the treatment regimens in a phase III setting.

DETAILED DESCRIPTION:
Once it is confirmed that the subjects fulfil the eligibility criteria and have signed the informed consent, they will be randomised to receive treatment based on cabazitaxel or vinflunine according to the following study schema:

(Randomize 1:1)

* Cabazitaxel 25 mg/m2 q3w
* Vinflunine 250-320 mg/m2 q3w

Random assignment of treatment will be stratified by the presence of 0 versus 1 of the following unfavourable prognostic risk factors proposed recently by Bellmunt et al. (1):

* Eastern Cooperative Oncology Group (ECOG) PS 1.
* Anaemia with Hb <10 g/dL.
* Presence of liver metastases.

All patients enrolled in the study will receive a cycle of treatment with the study medication (cabazitaxel or vinflunine) every 21 days until disease progression or intolerable/unacceptable toxicity. Tumour evaluations will be scheduled every 6 weeks until progression

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed TCCU (urinary bladder, urethra, ureter or renal pelvis). Patients with mixed histology may be enrolled if TCCU is the predominant component (i.e., > 50% of the histopathology sample) with the exception of neuroendocrine or small cell carcinoma.
* Advanced disease defined as a locally advanced tumour considered unresectable (T4b), node involvement in the inguinal area or above the aortic bifurcation (that are considered to be distant nodes and so metastasis) or metastasis in distant organs.
* Patient should have received one prior platinum-based chemotherapy treatment for locally advanced or stage IV TCCU. Prior platinum-based adjuvant or neoadjuvant therapy is allowed if more than 6 months have elapsed since the end of adjuvant or neoadjuvant therapy till tumour relapse.
* At least one measurable tumour lesion (measurable disease, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1
* ≥18 years.
* ECOG PS 0 or 1.
* May have no more than ONE of the following unfavourable risk factors:

  1. haemoglobin <10 g/dL
  2. presence of liver metastasis
  3. ECOG PS 1
* Life expectancy of at least 12 weeks.
* Adequate hematologic, hepatic, and renal function, defined by:
* Females of childbearing potential must have a negative serum pregnancy test within 7 days of study entry.

Exclusion Criteria:

* Patients that have 2 or more of the following unfavourable risk factors:

  1. Haemoglobin <10 g/L
  2. Liver metastasis
  3. ECOG PS 1.
* Women who are currently pregnant or breast-feeding.
* Any unresolved non-hematologic Adverse Event (AE) grade >1 (Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) Version 4.0) from previous anti-cancer therapy (other than alopecia)
* Patients who had undergone major surgery, radiation therapy or treatment with chemotherapy or any investigational agent within 28 days prior to Study day 1.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition
* History of another neoplasm.
* History of hypersensitivity reactions to taxanes (docetaxel) (cabazitaxel specific criteria), vinca alkaloids (vinflunine specific criteria) or to any of the formulation excipients, including polysorbate 80
* clear evidence or symptoms of central nervous system metastasis (cabazitaxel specific criteria).
* Clinically significant cardiac condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Phase II main objective: to assess the efficacy of cabazitaxel compared to vinflunine in terms of improved objective response rate (ORR) of subjects with metastatic or locally advanced previously treated TCCU. | From date of randomization to disease progression or until 18 months from enrolment.
  Efficacy of cabazitaxel compared to vinflunine on terms of improved objective response rate (ORR)
Phase III main objective: To assess the efficacy of cabazitaxel compared to vinflunine in terms of improved overall survival (OS) of subjects with metastatic or locally advanced, previously treated TCCU. | From date of randomization to death from any cause or until 18 months from enrolment.

SECONDARY OUTCOMES:
Phase II secondary objective: to assess the efficacy of cabazitaxel compared to vinflunine in terms of improved progression-free survival (PFS) and overall survival (OS). | From randomisation to either documented disease progression or death from any cause or until 18 months from enrolment (whichever occurs earlier)
Phase II secondary objective: safety profile and tolerability of cabazitaxel. It will be determined from the number of Adverse Events reported. | From the date the informed consent is signed up to 30 days after the last dose.
Phase III secondary objective: to assess the efficacy of cabazitaxel compared to vinflunine in terms of improved objetive response rate (ORR) and progression free survival (PFS). | From randomisation to either documented disease progression or death from any cause or until 18 months from enrolment (whichever occurs earlier)
Phase III secondary objective: safety profile and tolerability of cabazitaxel. It will be determined from the number of Adverse Events reported. | From the date the informed consent is signed up to 30 days after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt, MD/PhD, Principal Investigator — APRO
Locations (20):
- Netherlands (4):
  - NKI-AvL, Amsterdam, Amsterdam
  - Vumc Amsterdam, Amsterdam, Amsterdam
  - St. Antoniusziekenhuis, Nieuwegein, Nieuwegein
  - Erasmus MC Rotterdam, Rotterdam
- Spain (16):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Centro Oncologico de Galica, A Coruña, A Coruña
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Vall d´Hebron, Barcelona, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Morales Meseguer, Murcia, Murcia
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario Ourense. Hospital Santa María Nai, Ourense, Ourense
  - Hospital Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Lzoano Blesa, Zaragoza, Zaragoza

REFERENCES:
- [Background] Bellmunt J, Choueiri TK, Fougeray R, Schutz FA, Salhi Y, Winquist E, Culine S, von der Maase H, Vaughn DJ, Rosenberg JE. Prognostic factors in patients with advanced transitional cell carcinoma of the urothelial tract experiencing treatment failure with platinum-containing regimens. J Clin Oncol. 2010 Apr 10;28(11):1850-5. doi: 10.1200/JCO.2009.25.4599. Epub 2010 Mar 15. PMID 20231682
- [Derived] Bellmunt J, Kerst JM, Vazquez F, Morales-Barrera R, Grande E, Medina A, Gonzalez Graguera MB, Rubio G, Anido U, Fernandez Calvo O, Gonzalez-Billalabeitia E, Van den Eertwegh AJM, Pujol E, Perez-Gracia JL, Gonzalez Larriba JL, Collado R, Los M, Macia S, De Wit R; SOGUG and DUOS. A randomized phase II/III study of cabazitaxel versus vinflunine in metastatic or locally advanced transitional cell carcinoma of the urothelium (SECAVIN). Ann Oncol. 2017 Jul 1;28(7):1517-1522. doi: 10.1093/annonc/mdx186. PMID 28419193